CLINICAL TRIAL: NCT03553849
Title: Utilization of Very Low Calorie Diet in Obese General Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DDD603893 / 077069243
Record Dates: First submitted 2018-04-11; First posted 2018-06-12 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Morbid Obesity
Keywords: Very low calorie diet; General surgery
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Intervention Model Description: The patient will be randomized into the treatment or control arm by the research team. If they are randomized into the treatment arm, they will be prescribed with a 2-week VLCD that will begin 2 weeks prior to the scheduled elective surgery.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The operative surgeons will be blinded to the randomization. The patient, by nature of the study, will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Very Low Calorie Diet (Experimental): If they are randomized into the treatment arm, they will be prescribed with a 2-week VLCD that will begin 2 weeks prior to the scheduled elective surgery. Patients will be required to pay for the meal replacements.
  Interventions: Dietary Supplement: Very low calorie diet
- Standard Preop Diet (No Intervention): The control group will continue a regular diet until the day before surgery.

INTERVENTIONS:
Dietary Supplement: Very low calorie diet — The VLCD is a prescribed diet with well-balanced macro and micronutrients. It is intended for significant weight loss in a short period of time, is intended only for the extremely obese, and must be completed under the supervision of a trained physician.
  Arms: Very Low Calorie Diet

SUMMARY:
The investigators are studying the use of a two-week very low calorie diet (VLCD) in obese general surgery patients in a randomized single-blinded trial. The investigators hypothesize that the VLCD will positively impact the perceived surgical difficulty, operative time, hospital length of stay and 30-day complications. Additionally, the investigators anticipate reduced perioperative blood glucose levels and a reduced need for perioperative insulin administration.

DETAILED DESCRIPTION:
The investigators' objective for this project is to determine the impact of a preoperative VLCD on outcomes for patients undergoing elective general surgery. Included are patients who are obese, BMI >30, and scheduled by a Christiana Care-employed general surgeon for elective general surgery. Eligible patients are those scheduled for elective cholecystectomy, ventral or incisional hernia, umbilical hernia, and inguinal hernia surgery.

The investigators will also be determining the feasibility of introducing a preoperative VLCD for patients undergoing elective general surgery in a Community Hospital setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are obese, BMI >30, and scheduled by a Christiana Care-employed general surgeon for elective general surgery.
* Patients between the ages of 18 and 65.
* Patients scheduled for elective cholecystectomy, ventral or incisional hernia, umbilical hernia, and inguinal hernia surgery.

Exclusion Criteria:

* Patients will be excluded from the study if they have any of the following:

  1. Recent myocardial infarction (3-6 months).
  2. History of cerebral vascular accident (stroke).
  3. Diabetes mellitus with a history of severe ketoacidosis.
  4. Patients on SGLT2 inhibitors (glifozins) without insulin
  5. Chronic use of steroids, greater than 20mg daily.
  6. Bleeding peptic ulcer (unless there is radiological evidence of healing 6 months prior to entry).
  7. A psychiatric history that includes suicide attempts and anyone taking psychotropic drugs, including lithium carbonate.
  8. Active thrombophlebitis (or any other condition where decreased blood volume would put the patient at risk).
* In addition, patients who are pregnant are excluded. If status is unknown, a pregnancy test will be required prior to the start of the VLCD.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Reduction in Post Operative Complications | 30-days post operatively
  Pulmonary, cardiac and surgical complications using data collected from inpatient and outpatient charting

SECONDARY OUTCOMES:
Feasibility of the Study | 2 weeks
  Patient satisfaction and compliance based on patient surveys administered prior to discharge from the hospital
Effect on Perioperative BMI | 2 weeks
  Difference in pre operative and perioperative BMI, in kg/m^2
Effect on blood glucose levels | 2 weeks
  Difference in pre operative and perioperative blood glucose levels
Effect on insulin administration | 2 weeks
  Difference in pre operative and perioperative insulin administration, in units
Effect on operative times | Day of surgery
  Comparative operative times, in minutes, between control and intervention
Effect on operative blood loss | Day of surgery
  Comparative operative blood loss, in milliliters, between control and intervention
Effect on surgeon perceived difficulty | Day of surgery
  Comparative surgeon perceived difficulty between control and intervention utilizing a surgeon and procedure specific survey

CONTACTS AND LOCATIONS:
Overall Officials: Caitlin A Halbert, DO, MS, Principal Investigator — Christiana Care Health Services
Locations (1):
- Christiana Care Health System, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No